CLINICAL TRIAL: NCT03204682
Title: Repetitive Transcranial Magnetic Stimulation as an Analgesic Treatment in Endometriosis Chronic Pain : Feasibility Study
Brief Title: Repetitive Transcranial Magnetic Stimulation as an Analgesic Treatment in Endometriosis Chronic Pain : Feasibility
Acronym: ENDOSTIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-341; 2015-A01371-48 (Other: 2015-A01371-48)
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Deep Endometriosis; Chronic Pelvic Pain
Keywords: Endometriosis; Magnetic transcranial stimulation; Chronic pain; Analgesic
MeSH Terms: conditions — Endometriosis; Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants receive the same intervention throughout the protocol
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with chronic refractory endometriosis pain (Experimental): The aim of the study is to evaluate the feasibility of transcranial magnetic stimulation (rTMS) for analgesia on chronic refractory endometriosis pain.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Realization of a brain and medullary MRI to allow neuronavigation. Realization of 5 sessions of rTMS in 5 days during the first week then evaluation (physical examination, questionnaires) in consultation on post-stimulation. Then followed for 28 days in total through self-assessment of pain that will be filled daily on REDCap and last consultation on D28 for further evaluation

SUMMARY:
Endometriosis is associated with different types of pain (acute, chronic, excess nociception, neuropathic) generated by different mechanisms in the nervous system. The rTMS could provide significant analgesia for refractory endometriosis pain.

The aim of the study is to evaluate the feasibility of transcranial magnetic stimulation (rTMS) for analgesia on chronic refractory endometriosis pain.

DETAILED DESCRIPTION:
The first step consists of the inclusion of 12 patients followed by the filling by each patient of the RedCap software of five simple numerical scales for 4 weeks . Realization of a brain and medullary MRI to allow neuronavigation. Realization of 5 sessions of rTMS in 5 days during the first week then evaluation (physical examination, questionnaires) in consultation on post-stimulation. Then followed for 28 days in total through self-assessment of pain that will be filled daily on REDCap and last consultation on D28 for further evaluation

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal (presence of at least one of the two ovaries and absence of clinical signs of menopause),
* Not pregnant or breastfeeding;
* At least one painful symptoms related to the existence of endometriosis (dyspareunia, dysmenorrhea, pain with defecation or urination, neuropathic pain);
* Average VAS> 4/10, at least 4 days out of 7 for at least 3 months;
* Hormonal treatment failure continued in association or not for pain control;
* A level of understanding and satisfying expression in French;
* Monitoring possible during the duration of the study (4 weeks).
* These patients should be affiliated to the French social security and should have signed a written consent after receiving clear information.

Exclusion Criteria:

* Prior treatment with rTMS,
* Industrial accident or notion of litigation
* Cons-indication for rTMS (cortical lesion within 2cm of the motor cortex, ECT treatment during previous month, epilepsy and / or a history of epilepsy, history of head trauma, intracranial hypertension;
* Metal clip; pacemaker,
* Pregnant or breastfeeding women;
* Pain lasting less than 3 months;
* Another pain more severe than that associated with endometriosis;
* Lack of filling of the computerized questionnaires on Redcap;
* Incapable of understanding about informed consent,
* Patient under guardianship.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-04-13 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients tolerant 5 sessions of stimulation and with no increase in pain | at day 8
  The feasibility of rTMS treatment was defined if 7 patients or more over 12 tolerate the 5 sessions of stimulation showed no increase in pain

SECONDARY OUTCOMES:
Change in pain between the mean pain evaluated before inclusion | at day 8
  thanks to the visual analogue scale traded between 0 and 100
Endometriosis Health Profile Questionnaire (EPH-30); | at day 8
  Variation in scores of questionnaires before and after stimulation
Brief Pain Inventory (BPI): digital | at day 8
  Variation in scores of questionnaires before and after stimulation
Beck Questionnaire (Depression) | at day 8
  Variation in scores of questionnaires before and after stimulation
STAI of Anxiety Scale; Scale of alexythymie of Toronto | at day 8
  Variation in scores of questionnaires before and after stimulation
Catastrophizing Pain Scale (personality) | at day 8
  Variation in scores of questionnaires before and after stimulation
Quality of Life Questionnaire SF-36 | at day 8
  Variation in scores of questionnaires before and after stimulation
Migraine criteria (ICHD3) | at day 8
  Variation in scores of questionnaires before and after stimulation
Gastrointestinal quality of Life Index (GICLI) | at day 8
  Variation in scores of questionnaires before and after stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOURDEL, PH, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, Auvergne, France